CLINICAL TRIAL: NCT03446118
Title: Assessment of Fibrotic and Inflammatory Components by MRI in Strictures Associated With Eosinophilic Esophagitis Before and After Treatment
Brief Title: MRI to Assess Fibrosis in Eosinophilic Esophagitis Patients
Acronym: EoE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to lack of funding
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jeff Fidler, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17-006566
Record Dates: First submitted 2017-12-27; First posted 2018-02-26 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Eosinophilic Esophagitis
Keywords: EoE
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Intervention Model Description: Twenty patients with eosinophilic esophagitis will be studied. Ten of these patients will have mild to moderate stricture formation (narrowed segment <8 cm in length and lumen diameter > 12mm) and 10 will have small caliber esophagus (a narrowed segment >8 cm in length with minimum diameter < 10mm). These groups will be delineated by routine barium esophagography performed in all Mayo patients with eosinophilic esophagitis during their initial clinical evaluation. Patients will then undergo an 8 week treatment with 3 mg budesonide twice daily as per routine clinical treatment with clinically indicated follow up endoscopy with esophageal biopsies to assess mucosal response. All patients will complete the EESAI dysphagia score per routine practice at Mayo. MRI of the esophagus will be performed in these patients initially and upon completion of the 8 week course of steroid therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI to detect inflammation and fibrosis in EoE patients (Experimental): To assess through MRI the existence of an inflammatory and fibrotic component in strictures of eosinophilic esophagitis patients and to determine if this component is responsive to a therapeutic course of budesonide.
  Interventions: Diagnostic Test: MRI to detect inflammation and fibrosis in subjects with EoE

INTERVENTIONS:
Diagnostic Test: MRI to detect inflammation and fibrosis in subjects with EoE — MRI will be performed on a 1.5T magnet. Patients will be scanned in an oblique prone position similar to how esophageal distention is assessed at barium fluoroscopy

SUMMARY:
Can an MRI detect and monitor the inflammatory and fibrotic possess in patients with Eosinophilic Esophagitis

DETAILED DESCRIPTION:
MRI will be performed on a 1.5T magnet. Patients will be scanned in an oblique prone position similar to how esophageal distention is assessed at barium fluoroscopy. The following sequences and rationale will be used for the examination:

A sagittal 50mm thick multiphase FIESTA and multiphase SSFSE will be performed while the patient drinks water. The temporal resolution of the images will be approximately 1 image every 1.5-2 seconds. The images will be used to assess the lumen caliber and the wall thickness during maximal distension as pseudothickening can occur with decreased luminal distension.

Sagittal SSFSE with fat suppression, sagittal FRFSE T2-weighted images with fat suppression, axial DWI and sagittal DWI will be performed to asses for edema and inflammation within the esophageal wall.

axial FS SSFSE or FIESTA will be performed and targeted to the region of stricturing.

Dynamic sagittal imaging will be performed following IV contrast to assess for mural hyperenhancement which can be seen mural inflammation and delayed enhancement which can be seen in fibrosis. Sequential acquisitions will be performed beginning at 40 seconds following IV contrast injection. Delayed acquisitions will be performed at 5 min and 7 min. Patients will be asked to perform swallowing during the image acquisition to reduce the potential for pseudoenhancement secondary to under distension.

ELIGIBILITY:
Inclusion criteria:

* Adults ages 18-70 years of age
* Diagnosis of EoE, i.e. symptoms of esophageal dysfunction with histologic finding of 15 or more eosinophils per high power field on esophageal biopsy despite 8 weeks of high dose proton pump inhibitor therapy.
* All Subjects diagnosed with Eosinophilic Esophagitis pre and pose therapy

Exclusion criteria:

* Clinical evidence of infectious process potentially contributing to dysphagia (e.g. candidiasis, CMV, herpes)
* Other cause of dysphagia identified at endoscopy or esophagram (e.g. reflux esophagitis, stricture, web, ring, achalasia, esophageal neoplasm)
* Esophageal minimal diameter < 13 mm on structured barium esophagram
* Inability to read due to: Blindness, cognitive dysfunction, or English language illiteracy
* Pregnant women
* Presence of body metallic fragments or devices that prohibit use of MRI
* History of renal disease
* eGRF <30

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Measurement of distinct inflammatory and fibrotic components of the esophageal stricture in patients with eosinophilic esophagitis | 1 day
  At 5,15 and 25 cm above the gastroesophageal junction and in areas of obvious esophageal thickness, digitized areas of inflammation and fibrosis will be measured individually and as a proportion of overall esophageal diameter in that area before and after steroid treatment.

SECONDARY OUTCOMES:
Barium Esophagram | 1 day
  The barium esophagram will measure moderate stricture formation to delineate the groups- Group 1.(narrowed segment <8 cm in length and lumen diameter > 12mm) and Group 2- 10 will have small caliber esophagus (a narrowed segment >8 cm in length with minimum diameter < 10mm).
Eosinophilic Esophagitis Activity Index (EEsAI) | 1 day
  Questionnaire developed to measure dysphagia - using the pro scoring method

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Fidler, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials